CLINICAL TRIAL: NCT04135625
Title: Improving Nutrition in Children Under Two Through Increased Egg Consumption in Burkina Faso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB201702810; AID-OAA-L-15-00003 (Other Grant/Funding Number: US AGCY INTL DEV)
Record Dates: First submitted 2019-10-11; First posted 2019-10-22 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Nutrition
MeSH Terms: interventions — alpha-internexin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Control Group - with no chickens gifted and no INA training sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full Intervention (Active Comparator): The full intervention group will receive three egg laying chickens that will be presented as a gift to the child by their religious leader (imam or priest) during a gifting ceremony, as well as Integrated nutrition and agricultural (INA) education training sessions.
  Interventions: Behavioral: Integrated nutrition and agricultural (INA) trainings; Behavioral: Ceremonial Gifting of Livestock
- Education Only (Active Comparator): The education only intervention group will receive 3 chickens given in manner similar to animal distribution programs and the INA training sessions.
  Interventions: Behavioral: Integrated nutrition and agricultural (INA) trainings
- Control (No Intervention): The control group will receive no chickens gifted and no INA training sessions.

INTERVENTIONS:
Behavioral: Integrated nutrition and agricultural (INA) trainings — Monthly INA training session to help increase knowledge about nutrition and chicken husbandry and help to increase resiliency on a household level.
  Arms: Education Only; Full Intervention
Behavioral: Ceremonial Gifting of Livestock — Egg laying chickens will be presented as a gift to the child by a community champion (their religious leader or village chief)) during a gifting ceremony
  Arms: Full Intervention

SUMMARY:
This project targets vulnerable populations of smallholders, women and children and should lead to increased poultry production, increased egg consumption of children, improved nutrition, and increased household level resilience. This innovative intervention will be the gifting of chickens by religious leaders to children ages 6 to 12 months coupled with integrated nutrition and agricultural trainings.

DETAILED DESCRIPTION:
This study involves innovative behavioral change theoretical methodology to empower caregivers as smallholder poultry producers by improving their access to livestock production resources and agricultural extension services, providing tools for improved decision making, and enhancing nutrition based knowledge. Smallholder production is important in eliminating food insecurities and building resilience to improve nutrition in children under 5. Based on the results of the Ethiopian egg project, through messaging and education, this study will foster favorable attitudes and consequent behavioral changes, including increased egg consumption.

ELIGIBILITY:
The study population will be selected with the assistance of the OCADES Caritas Kaya and the CHWs who are actively involved and trusted within the targeted village communities.

Inclusion Criteria:

* Living within the identified areas of the study population

Exclusion Criteria:

* history of egg allergies
* severe malnutrition

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Increase egg consumption in children under two living in Kaya, Burkina Faso | Baseline up to 12 months
  Dietary recall survey requesting caregiver/ parental recall of their child's dietary intake over the past week to include egg consumption embedded within the questionnaire The percentage of children consuming eggs will be calculated based on a yes response from the parent.The outcome measure will be described as the percentage of children consuming eggs with in the study population.
Increase egg consumption frequency in children under two living in Kaya, Burkina Faso | Baseline up to 12 months
  Dietary recall survey requesting caregiver/ parental recall of their child's dietary intake over the past week to include frequency of eggs given embedded within the questionnaire.The outcome measure will be described as the mean number of eggs consumed in the past week by children enrolled in the study that consume eggs .

SECONDARY OUTCOMES:
Improve growth in children under two living in Kaya, Burkina Faso. | Baseline up to 12 months
  Anthropometric measurements to include weight in kilograms, height in centimeters of enrolled children. Measurements will be aggregated to calculate z scores based on the child's age calculated in days and the wight and height of the anthropometric measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah McKune, PhD, MPH, Principal Investigator — University of Florida
Locations (1):
- Institut de l'Environnement et Recherches Agricoles (INERA), Ouagadougou, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared on a USAID data development library and DataVerse.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be shared with six months time completion. USAID will review and determine the level of access.
  IPD uploaded to Dataverse.
Access Criteria: USAID will review and determine the level of access and the time length the data is shared. Data uploaded to DataVerse will be available indefinitely.
URL: https://dataverse.harvard.edu/dataverse/livestock-lab-burkina-egg-consumption .

REFERENCES:
- [Derived] McKune SL, Stark H, Sapp AC, Yang Y, Slanzi CM, Moore EV, Omer A, Wereme N'Diaye A. Behavior Change, Egg Consumption, and Child Nutrition: A Cluster Randomized Controlled Trial. Pediatrics. 2020 Dec;146(6):e2020007930. doi: 10.1542/peds.2020-007930. PMID 33239474
- [Derived] Stark H, Omer A, Wereme N'Diaye A, Sapp AC, Moore EV, McKune SL. The Un Oeuf study: Design, methods and baseline data from a cluster randomised controlled trial to increase child egg consumption in Burkina Faso. Matern Child Nutr. 2021 Jan;17(1):e13069. doi: 10.1111/mcn.13069. Epub 2020 Aug 8. PMID 32770664